CLINICAL TRIAL: NCT01994967
Title: Study Phase III to Evaluate the Noninferiority of Heavy Levobupivacaine 50% Enantiomeric Excess (Levobupivacaine S75:R25) Compared to Racemic Heavy Bupivacaine (Bupivacaine S50:R50) in Spinal Anesthesia for Lower Limb Orthopedic Procedures
Brief Title: Phase III, Evaluate Noninferiority Between Levobupivacaine and Bupivacaine in Spinal Anesthesia.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Another regulatory way was defined.
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Collaborators: Newco Trials Pesquisa Científica Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRT074
Record Dates: First submitted 2013-10-30; First posted 2013-11-26 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Orthopedic Disorder of Spine
Keywords: Phase III; Noninferiority; Controlled; Double-blind; Randomized; Spinal; Anesthetic; Lower limb
MeSH Terms: interventions — Levobupivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levobupivacaine (Experimental): Presentation: injectable solution - ampoule of Levobupivacaine Hydrochloride
  Indication: production of subarachnoid block (spinal/ spinal anesthesia).
  Interventions: Drug: Levobupivacaine
- Bupivacaine (Active Comparator): Presentation: injectable solution - ampoule of Bupivacaine Hydrochloride
  Indication: production of subarachnoid block (spinal/ spinal anesthesia).
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — Will be administered 3 ml of the investigational anesthetic in combination with morphine through the subarachnoid via.
  Other Names: Levobupivacaine Hydrochloride.
  Arms: Levobupivacaine
Drug: Bupivacaine — Will be administered 3 ml of the investigational anesthetic in combination with morphine through the subarachnoid via.
  Other Names: Neocaína ®.; Bupivacaine Hydrochloride.
  Arms: Bupivacaine

SUMMARY:
Clinical trial phase III, noninferiority, controlled, double-blind, randomized. The purpose of this study is to evaluate the noninferiority between Levobupivacaine and Bupivacaine in spinal anesthesia.

DETAILED DESCRIPTION:
Objectives:

Primary:

* Evaluation of latency to sensory block of T10.
* Evaluation of the duration of sensory block.

Secondary:

* Evaluation of the motor block degree.
* Evaluation of motor block duration.
* Evaluation of cardiovascular safety.
* Block failure.
* Observation of adverse events.

Study Plan:

* Estimated 120 research participants;
* Aged between 18 - 80 in both gender;
* Drug Intervention: 01 day

Evaluations during Trial:

* Classification of anesthetic risk: Class I to VI by the American Society of Anesthesiologists(ASA);
* Identification of the Anesthetic Failure;
* Latency time for sensory block at T10;
* Duration of sensory block and motor block;
* Bromage scale;
* Cardiovascular safety;

Retention of Records:

The investigator shall retain all documentation of the study over a period of at least five years from the end of the study. The Sponsor or its designee will provide a list of all documentation which should be kept by the Investigator.

Monitoring:

All aspects of the study will be carefully monitored by Cristália Pharmaceutical Chemicals Ltda. or designated representative of it (Clinical Research Organization - CRO) for evaluations related to good clinical practice and applicable local regulations.

Case Report Forms. The Monitor will be available if the investigator, or other person of his team, needs information and guidance.

The Monitor of the study should have permanent access to all documentation and it is his obligation to ensure that the Case Report Forms are complete and completed correctly, as well as checking if the data are described according to the source documents, in order to eliminate interferences that may compromise the accuracy of the data generated in the clinical trial.

Audit and Inspections:

Authorized representatives of the Sponsor or designees, regulatory authority or the Ethics Committee of the institution may conduct audits or inspections during or after the study conclusion.

Collecting Data:

The information corresponding to the data of interest from the study will be collected and recorded in Case Report forms provided by Sponsor, and filled from the information contained in the source documents.

Documents are considered sources for study: medical records used by the professional at the time of the visits, diagnostic tests or image.

Informed Consent of Trial:

The Principal Investigator will ensure that the research participant receive verbally and in writing all relevant information about the nature, purpose, the test drug, the possible risks and benefits of the study.

Research participants will be notified that they are free to discontinue the study at any time. That they will have the opportunity to ask questions and to have sufficient time to consider the information received.

Formation of the database:

The database of the study will be assembled with the data from the Case Report Forms. Doubts and discrepancies will generate questions (queries) written to the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes;
* Age between 18 and 80 years;
* Risk anesthetic classified as ASA I or ASA II, according to the American Society of Anesthesiology;
* What have indication for spinal orthopedic surgery in the lower limbs;
* Have agreed to participate and signed the informed consent form.

Exclusion Criteria:

* Absolute or relative contraindications to spinal anesthesia;
* Hypersensitivity or intolerance to local anesthetics or to components of the formula;
* Spinal cord injuries, peripheral neuropathy or other neurological condition that lead to sensitivity and/ or motor function disorder;
* Dementia, mental retardation and others important cognitive changes;
* Obesity with a body mass index ( BMI ) ≥ 35 or difficulty in executing the puncture;
* Anatomical column difficulty in the opinion of the investigator;
* Previous spine surgical intervention;
* Polytrauma;
* Tattoo at the puncture site;
* Alcoholism;
* Abuse of illicit substances;
* Antecedents of severe anaphylactic reactions or Steven - Johnson disease;
* Changes in security checks;
* Participation in a clinical study in the 12 months preceding this inclusion;
* Pregnancy and lactation;
* Any other condition that in the opinion of the investigator, may lead to increased risk for the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Time of latency to achieve sensitive block of T10. | 01 day.
  The interval of time between the withdrawal of the needle at the end of local anesthetic injection and the absence of response to sensory stimulus in the region corresponding to the T10.
Duration time of the sensory block of T10. | 01 day.
  Duration of anesthesia as for the sensory aspect through a needle stimulus in the anterior side of the foot.

SECONDARY OUTCOMES:
Sensory block intensity. | 02 days.
  Ability of the patient to move their lower limbs, assessed by Bromage scale.
Motor block duration. | 02 days.
  Time interval between the end of anesthetic injection and the return to 0 score in modified Bromage scale.
Cardiovascular safety. | 02 days.
  Incidence and severity of hemodynamic (BP and HR) and respiratory (SpO2) alterations.
Block failure. | 02 days.
  To evaluate the absence of signs of analgesia or motor block for at least 20 minutes after anesthetic injection in the sensitive region studied.
Adverse events. | 02 days.
  To evaluate the occurrence of adverse events regarding the frequency, duration, severity and causal relationship with the study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Onésimo D. Ribeiro Junior, Medic, Principal Investigator — CEMEC
Locations (5):
- Brazil (5):
  - IMIP - Instituto de Medicina Integral Prof. Fernando Figueira, Recife, Pernambuco
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Hospital de Base de São José do Rio Preto /SP, São José do Rio Preto, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da USP / SP, São Paulo, São Paulo
  - CEMEC - Multidisciplinary Center of Clinical Studies, São Paulo